CLINICAL TRIAL: NCT03348865
Title: Interventions to Reduce Psychological Interventions Associated With Infertility in Nigeria.
Brief Title: Fertility Life Counselling Aid- FeLiCiA
Acronym: FeLiCiA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Weeks MD MRCOG (Other)
Collaborators: University of Liverpool (Other); University College Hospital, Ibadan, Nigeria (Unknown)
Responsible Party: Sponsor-Investigator, Andrew Weeks MD MRCOG, Professor of International Maternal Health, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2121
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Infertility/Sterility; Psychological Distress; Psychological Stress; Anxiety Disorders; Depressive Disorder
Keywords: Cognitive Behavioural Therapy
MeSH Terms: conditions — Infertility; Stress, Psychological; Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fertility Life Counselling Aid (FeLiCiA) (Experimental): Patients to undergo weekly Felicia counselling interventions for 6 weeks; making a total of 6 sessions.
  Each session is expected lasts 30 mins to 1 hour.
  Interventions: Behavioral: Fertility Life Counselling Aid (FeLiCiA)
- Control (No Intervention): Patients are to undergo treatment as usual.

INTERVENTIONS:
Behavioral: Fertility Life Counselling Aid (FeLiCiA) — The FeLiCiA study is a pilot randomised control trial study of an intervention that uses cognitive behavioral therapy (CBT) method to provide counselling for infertility patients within low resource settings. this intervention is designed for management of the psychological problems associated with having infertility. It is based on the Thinking Healthy Programme by WHO.
  Arms: Fertility Life Counselling Aid (FeLiCiA)

SUMMARY:
Research Objectives:

1. To test the FeLiCiA, a 6 week intervention developed for the management of psychological morbidities associated with infertility, using external randomised control trial methods, on patients showing positive indicators for psychological morbidity amongst patients with infertility at UCH Ibadan, Nigeria.
2. To explore and understand patient perspectives on the benefits of the FeLiCiA counselling in addition to usual clinical care.

Summary of Research:

Population:

Sample size N=42 Men & Women (aged 21-45) with GHQ 12 score indicative of mild to moderate psychological morbidities (3 or more) among patients attending University College Hospital for infertility treatment.

Intervention:

FELICIA [N= 21 intervention] 6 weekly counselling Follow up at 6/52 and 6/12. Inclusion Criteria: Age 21-45; Exclusion Criteria: Previously diagnosed mental illness; severe anxiety & depression or suicide intent (immediate referral); Age<21/>45.

Comparison: [N=21 control group] Treatment as usual

Outcome:

Primary-GHQ12 score less than 3 Secondary-

1. Sustained GHQ12 score less than 3
2. Patient perspectives on benefits and effectiveness of intervention, and patient empowerment post intervention.

DETAILED DESCRIPTION:
Eligible participants will be recruited by randomisation into a pilot trial of the intervention. The pilot trial will be in two groups- the intervention group (FELICIA) and the control group (No intervention/ treatment as usual). The intervention group will be see undergo a 6 weekly counselling sessions, using the FELICIA manual to deliver infertility counselling. The counselling sessions are to be delivered by the nurses at the infertility clinic who will be trained by the researcher to deliver this intervention. The FeLiCiA manual was developed by Dr Abiola Aiyenigba who is the principal investigator. FeLiCiA is based on the THINKING HEALTH PROGRAMME developed by Prof Atif Rahman, who will also be supervising the research. Further details are available in the FeLiCiA manual, which is attached to his proposal for further reference.

Semi structure interviews: Qualitative research will be carried out using one to one interviews. Patient will be asked to discuss their views regarding the benefits of the intervention in helping them manage the stresses that they face dealing with infertility.

Study Site:

The study will be carried in the University College Hospital, Ibadan, Nigeria Study Population The study population will consist of patients attending clinics for the treatment of infertility at the University College Hospital, Ibadan, Nigeria

Sampling Method (N=42):

For the external pilot RCT for testing the FeLiCiA intervention, thirty-eight patients are required to have an 80% chance of detecting, as significant at 5% level, an increase in the primary outcome measure from 5% in the control group to 40% in the experimental group. We increase this sample size by 10% to account for drop out during the 6 weeks, making up a total of 42 patients to be recruited for the trial.

Randomization:

The participants who have consented to participate in the research will be randomized into 2 groups - the Intervention group and the Control Group. The randomization is blinded and allocated using sealed opaque envelopes. The envelopes have been prepared by an independent person; all those carrying out the research have no idea what the contents of the envelopes indicate.

Patients who are eligible and wish to continue with the research will be handed a brown sealed envelope, opened for the first time in the presence of the participant. Depending on the content of the envelope patients will be randomized into either the intervention or control group.

The intervention group will receive the FeLiCiA counselling intervention while the Control group will receive treatment as usual. Counselling sessions will take place via discussion once every week for six weeks. Each counselling session will last no more than 1 hour. Interviews will also take place at the 2 follow up periods at the end of the sis weeks counselling and six months post counselling. (See follow up procedure).

Semi structure interviews:

Participants recruited for the qualitative study (one to one interviews) will be interviewed on one occasion for one to one qualitative research. An interview sessions is expected to last no more than 1 hour.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting Patients aged between 21 and 45 years attending the infertility outpatient clinics, the Assisted Reproduction clinics and other gynecological, andrology and nephrology clinics for infertility treatment
2. Patients who have been undergoing infertility treatments for over 2 years.
3. Patients who also have a GHQ 12 score of 3 or more.
4. Patients who have been identified having mild to moderate anxiety and/or depression using the psychometric measuring tools that would not qualify to be treated bio-medically.

Exclusion Criteria:

1. Non-consenting patients aged between 21 and 45 years attending the infertility outpatient clinics, the Assisted Reproduction clinics and other gynecological, andrology and nephrology clinics for infertility treatment.
2. Participants with infertility for less than two years.
3. Participants identified as having severe forms of anxiety and depression that require urgent psychiatric treatments/referral.
4. Patients who have previously been clinically diagnosed and treated for with a mental illness.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement for absence of psychological morbidities post intervention | 6 weeks
  GHQ 12 score= less than 3 - No psychological morbidities

SECONDARY OUTCOMES:
Explore patient perspective on benefits of intervention using qualitative methods, post intervention. | 6 weeks
  One to one semi structured interviews to gain patient perspectives on 1. benefits of intervention, and 2. Patient feelings of empowerment post intervention
Measurement for sustained absence of psychological morbidities, 6months post intervention | 6 months
  GHQ 12 score= less than 3 - No psychological morbidities

CONTACTS AND LOCATIONS:
Overall Officials: Abiola O Aiyenigba, PhD Student, Principal Investigator — University of Liverpool
Locations (1):
- University College Hospital, Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided